CLINICAL TRIAL: NCT04789044
Title: A Phase 2a Multicenter Randomized Controlled Trial Evaluating the Safety and Efficacy of Polyethylene Glycol (PEG) Mediated Fusion (PEG Fusion) Compared to Standard of Care in the Repair of Mixed Motor-sensory Acute Peripheral Nerve Injuries (PNI) for Rapid and Immediate Improvement in Outcome
Brief Title: Evaluating the Safety and Efficacy of Polyethylene Glycol (PEG) Mediated Fusion (PEG Fusion)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH2010825
Record Dates: First submitted 2021-02-22; First posted 2021-03-09 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Intervention Model Description: The study will enroll 40 patients receiving autograft reconstruction within 24 hours of injury. Patients within each group will be randomized to either PEG mediated reconstruction (n=20); or conventional nerve reconstruction (n=20).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEG mediated reconstruction (Experimental): NTX-001 will be administered topically via isolation chamber medical device. Dose Unit: 2.5 mL NTX-001 is a single use surgical product intended for use as adjunct treatment in the repair of severed peripheral nerves in patients requiring standard suture neurorrhaphy.
  Interventions: Drug: NTX-001
- Conventional nerve reconstruction (No Intervention): Conventional nerve reconstruction

INTERVENTIONS:
Drug: NTX-001 — • PEG fusion is the application of a polyethylene glycol (PEG) using a combination of sequenced reagents to a freshly performed nerve coaptation, or neurorrhaphy, to allow the axonal membranes of the proximal and distal axonal stumps to fuse back together and re-establish full axonal continuity.
  Arms: PEG mediated reconstruction

SUMMARY:
The overall objective of this study is to determine the safety of PEG fusion when used with primary repair or reconstruction in patients with an acute upper extremity peripheral nerve injury. PEG is safe and effective for extending the half-life of circulating pharmaceutical products, when used in conjunction with a topical hemostatic agent in surgical wounds, and when used as a colon cleanser for endoscopic surgical procedures. However, PEG fusion has not been rigorously tested as a safe reagent to promote nerve regeneration in humans. Therefore, the goal of this Phase 2a clinical trial is to establish safety data and to examine the effect of PEG fusion on clinical outcomes including recovery of sensory and motor function. Results will be externally validated using data collected in the DoD funded prospective NERVE study and will provide preliminary evidence to power a larger phase II efficacy trial.

DETAILED DESCRIPTION:
The study will enroll 40 patients receiving autograft reconstruction within 24 hours of injury. Patients will be randomized to either PEG mediated reconstruction (n=20); or conventional nerve reconstruction (n=20). The investigators hypothesize that (1) the rate of complications within 1 month of surgery in patients treated with PEG fusion will be comparable to that of patients treated with conventional autograft reconstruction, (2) there will be no detrimental effects from PEG fusion on nerve regeneration over 2 years compared to patients treated with conventional nerve reconstruction, ((3) recovery of sensory and motor function will occur earlier (within 6 months) among patients treated with PEG fusion compared to patients treated with conventional autograft reconstruction (4) patients treated with PEG fusion will have better range of motion, greater hand strength, less disability, less pain, and higher rates of treatment satisfaction compared with patients treated with conventional autograft reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-80
2. Sustained a complete peripheral nerve injury resulting from upper extremity trauma presenting within 48 hours of injury
3. Involves injury or dysfunction to motor and/or sensory function of the axillary, radial, median, ulnar, or musculocutaneous nerve with injury localized between the proximal humerus and the distal flexion crease of the wrist
4. Involves a "mixed" nerve segment (i.e., involves a location of any of the above specified nerves that can be expected to have both sensory and motor axons present).

Exclusion Criteria:

1. Patients beginning surgery within hours after injury.
2. Injury to the brachial plexus nerves
3. Injury to the nerves distal to the distal flexion crease of the wrist
4. Injury that involves a distal extension of the parent nerve that is considered sensory only (superficial radial nerve, lateral antebrachial cutaneous nerve, etc.) or the posterior interosseus or anterior interosseus nerve distal to the midpoint of the forearm (i.e., distal to what can be considered the main motor branches of the PIN and AIN).
5. Previous peripheral nerve injury resulting from trauma, stroke, muscular, neurologic, or neuromuscular disorder
6. Documented psychiatric disorder that is expected to result in high probability of self-harm or interfere with study follow-up.
7. Severe problems with maintaining follow up (e.g., patients who are prisoners or homeless at time of injury or who are intellectually challenged without adequate family support).
8. Not expected to survive the next 30 days due to their injuries/health condition.
9. The subject has a known allergy to polyethylene glycol (PEG).
10. If any of the assessments cannot be done on the contralateral side (CL) or the MRCC sensory 2PD value is > 10 mm on the CL side during baseline period, the subject is a screen failure.
11. The subject is pregnant and/or is breastfeeding.
12. The subject has a significant medical comorbidity precluding immediate repair.
13. The subject is not able to strictly adhere to the rules of the current clinical protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Complications or problems that occur with in the first 30 days. | Up to 2 years
  Complications or problems include surgical site infections, wound dehiscence/breakdown, exposure of nerves and/or their repairs and reconstructions, breakdown of nerve repair or reconstruction, seroma/hematoma requiring an additional procedure to treat, and any other local wound complications related to the zone of nerve injury that require an additional surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie Shores, MD, Principal Investigator — Johns Hopkins University
Locations (7):
- United States (7):
  - University of Maryland Medical Center Shock Trauma Center, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - OrthoCarolina, Charlotte, North Carolina
  - Wellspan Health, York, Pennsylvania
  - San Antonio Military Medical Center (SAMMC), San Antonio, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No